CLINICAL TRIAL: NCT04867447
Title: Prevalence of Traumatic Events and Post-traumatic Stress Disorder in Immigrant and Non-immigrant Patients With Psychotic Disorder
Brief Title: Prevalence of Traumatic Events and PTSD in Immigrant and Non-immigrant Patients With Psychotic Disorder
Status: Completed | Type: Observational
Sponsor: Parc de Salut Mar (Other)
Collaborators: Universitat Autonoma de Barcelona (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/8398/I
Record Dates: First submitted 2021-04-12; First posted 2021-04-30 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-04

CONDITIONS: Psychotic Disorders; Psychological Trauma; Stress, Psychological; Cross-Cultural Comparison
MeSH Terms: conditions — Psychotic Disorders; Psychological Trauma; Stress, Psychological

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case-Immigrants psychotic patients: Individuals who have presented at least one non-affective psychotic episode with an immigrant status, defined as "a person who migrates to another country, usually for permanent residence"
  Interventions: Diagnostic Test: Psychological trauma evaluation
- Control-Non immigrants psychotic patients: Individuals who have presented at least one non-affective psychotic episode who do not have an immigrant status.
  Interventions: Diagnostic Test: Psychological trauma evaluation

INTERVENTIONS:
Diagnostic Test: Psychological trauma evaluation — Psychological trauma exposure is assessed by validated scales:
  * Childhood Trauma Questionnaire (CTQ)
  * Clinician-Administered PTSD Scale for DSM-5 (CAPS-5)
  * Cumulative Trauma Scale.
  * The Holmes and Rahe Stress Scale.
  Other clinical scales used:
  * Positive and Negative Syndrome Scale (PANSS).
  * Dissociative Experiences Scale (DES)
  * Mini-Mental State Examination (MMSE).

SUMMARY:
Higher rates of psychosis are described in migrant population. Likewise, this populations could suffer several adversities during migration process that could lead to higher exposure to traumatic events and higher rates of posttraumatic stress disorder (PTSD). There is a growing evidence that trauma is associated with psychosis onset.

The aim of this research is to study the association between psychosis and traumatic events exposure/PTSD in immigrant population. Our hypothesis is that the higher incidence of psychosis described in immigrant population is associated to higher trauma exposure.

A case-control observational study is performed. Patients who presented at least one psychotic episode are recruited from acute and chronic units at "Parc Salut Mar" (Barcelona). Estimated total sample is 196 individuals. Trauma exposure is assessed by validated trauma scales. Known factors associated with psychosis are controled during the statistic analysis.

ELIGIBILITY:
Inclusion Criteria:

* To present history of one or more psychotic episodes defined according to DSM-5 criteria, including patients with diagnoses of Schizophrenia, Schizoaffective Disorder and non-specific psychotic disorders.
* Patients of non-local origins who have undergone a migration process along the life line (as case individuals) and autochthonous patients (as control individuals).
* Age between 18 and 65 years.

Exclusion Criteria:

* Patients who have not clinical stability.
* Important cognitive limitations to understand informed consent nor applied questionnaires.
* Language barrier that limits understanding informed consent nor applied questionnaires.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present, according DSM-V criteria, one or more non-affective psychotic episodes from Acute and Chronic inpatients units at Parc de Salut Mar (Barcelona).
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Childhood Trauma exposure | From birth to age 18 (216 months)
  Assessed by Childhood Trauma Questionnaire (CTQ): is a self-administered 28-item scale to measure abuse and neglect suffered in childhood on five subscales: emotional, physical or sexual abuse, and emotional or physical neglect, each subscale scored on a 5-point Likert scale. The score for each subscale classifies the severity of the abuse and neglect as: "none to minimal," "low to moderate," "moderate to severe" and "severe to extreme".
Global Trauma exposure by Cumulative Trauma Scale | From birth to study evaluation, assessed up to 250 months.
  Cumulative Trauma Scale (CTS): Assesses exposure and emotional involvement to 33 traumatic events, especially oriented to minority groups such as refugees, prisoners or mental health patients. Each item on a 7-point Likert scale (from "1-extremely positive to 7-extremely negative"). Higher scores show more cumulative lifetime traumatic events exposure.
The Holmes and Rahe Stress Scale | 1 year (previous to study evaluation) .
  The Holmes and Rahe Stress Scale (Holmes & Rahe): is used to determine which common stressful life events a patient has experienced in the last 12 months, with each life event scored according to a standardized measure of their impact and a total score provided by summing all those applicable to the patient. Scores <150 are correlated with low stress, 150-299 scores are correlated with moderate stress and >300 scores are correlated with high level of stress.
PTSD prevalence | From birth to study evaluation, assessed up to 250 months.
  Clinician-Administered PTSD Scale for Diagnostic and statistical manual of mental disorders 5th edition (DSM-V), (CAPS-5): is a 55-item clinician-applied scale to determine PTSD diagnosis, based on the current DSM-V criteria. This scale consists of three sections: events, symptoms and functioning.

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | 1 week (previous to study evaluation)
  Psychotic symptoms are measured with the Positive and Negative Syndrome Scale (PANSS) for schizophrenia an 30-item clinician administered scale which measures positive, negative and general psychopathological symptoms on a scale of 1-7, based on the severity of the symptom (1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, and 7=extreme). The higher scores are correlated with more severe symptomatology.
  A total score of 58 indicates "moderate severity," while a PANSS score of 75 represents "marked severity." A PANSS total score of 95 corresponds to "severe severity," and a score of 116 signifies "very severe severity."
Dissociative symptoms prevalence | 1 week (previous to study evaluation)
  Dissociative Experiences Scale (DES): is a 28-item self-report scale which measures the frequency with which an individual experiences a range of dissociative experiences, from normal to pathological. An overall mean score ranges from 0 to 100, and there are subscales for amnesia, dissociation and depersonalization. A total score of over 30 indicate high levels of dissociation
Substance use disorder prevalence. | From birth to study evaluation, assessed up to 250 months.
  A diagnosis of substance use disorder (alcohol or other illicit substances) will be made according to Diagnostic and statistical manual of mental disorders 5th edition (DSM-V) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Amira Trabsa Biskri, MD, Principal Investigator — Institut Hospital del Mar d'Investigacions Mèdiques (IMIM)
Locations (1):
- Unidad de Investigación del Centro Fórum y Instituto Hospital del Mar de Investigaciones Médicas., Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Betancourt TS, Newnham EA, Birman D, Lee R, Ellis BH, Layne CM. Comparing Trauma Exposure, Mental Health Needs, and Service Utilization Across Clinical Samples of Refugee, Immigrant, and U.S.-Origin Children. J Trauma Stress. 2017 Jun;30(3):209-218. doi: 10.1002/jts.22186. Epub 2017 Jun 6. PMID 28585740
- [Result] Cantor-Graae E, Selten JP. Schizophrenia and migration: a meta-analysis and review. Am J Psychiatry. 2005 Jan;162(1):12-24. doi: 10.1176/appi.ajp.162.1.12. PMID 15625195
- [Result] Anderson KK, Edwards J. Age at migration and the risk of psychotic disorders: a systematic review and meta-analysis. Acta Psychiatr Scand. 2020 May;141(5):410-420. doi: 10.1111/acps.13147. Epub 2020 Jan 20. PMID 31903545
- [Result] Hollander AC, Dal H, Lewis G, Magnusson C, Kirkbride JB, Dalman C. Refugee migration and risk of schizophrenia and other non-affective psychoses: cohort study of 1.3 million people in Sweden. BMJ. 2016 Mar 15;352:i1030. doi: 10.1136/bmj.i1030. PMID 26979256
- [Result] Selten JP, Hoek HW. Does misdiagnosis explain the schizophrenia epidemic among immigrants from developing countries to Western Europe? Soc Psychiatry Psychiatr Epidemiol. 2008 Dec;43(12):937-9. doi: 10.1007/s00127-008-0390-5. No abstract available. PMID 18587677
- [Result] Gibson LE, Alloy LB, Ellman LM. Trauma and the psychosis spectrum: A review of symptom specificity and explanatory mechanisms. Clin Psychol Rev. 2016 Nov;49:92-105. doi: 10.1016/j.cpr.2016.08.003. Epub 2016 Aug 31. PMID 27632064
- [Result] Howes OD, McCutcheon R. Inflammation and the neural diathesis-stress hypothesis of schizophrenia: a reconceptualization. Transl Psychiatry. 2017 Feb 7;7(2):e1024. doi: 10.1038/tp.2016.278. PMID 28170004
- [Derived] Trabsa A, Redolar-Ripoll D, Vargas L, Llimona A, Hogg B, Valiente-Gomez A, Perez V, Moreno-Alcazar A, Amann BL. A comparison of PTSD and traumatic event rates in a clinical sample of non-refugee immigrants and native-born individuals with a psychotic disorder: a case-control study. Eur J Psychotraumatol. 2023;14(2):2263151. doi: 10.1080/20008066.2023.2263151. Epub 2023 Oct 17. PMID 37846737